CLINICAL TRIAL: NCT07068880
Title: Clinical Analysis of a Novel Flexor Tendon Repair Technique, A Prospective Randomized Trial
Brief Title: Clinical Analysis of a Novel Flexor Tendon Repair Technique
Status: Recruiting | Type: Observational
Sponsor: Brett Lewellyn (Other)
Responsible Party: Sponsor-Investigator, Brett Lewellyn, Chief Hand & Upper Extremity Surgery, Orlando Health, Inc.
Organization: Orlando Health, Inc. (Other)
Other Study IDs: 23.184.09
Record Dates: First submitted 2025-06-23; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Flexor Tendon Laceration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- repair with the CoNextions tendon repair device
- repair with a "standard of care" repair technique known as the Lew-Omar (LO) technique

SUMMARY:
The purpose of the research study is to determine the efficacy and efficiency of two tendon repair techniques: the CoNextions tendon repair device vs a standard of care, L-O (Lew-Omar), suture repair technique. The investigators will also determine if there are similar or different rates of complications and failures via both objective and subjective measures.

DETAILED DESCRIPTION:
To determine the tendon failure/rupture rate of two tendon repair techniques: the CoNextions tendon repair device vs a standard of care suture repair technique. The investigators will determine if there are similar or different rates of complications and failures (both intraoperatively and at 2-week, 6-week, 3-month, and 6-month post-operative intervals).

ELIGIBILITY:
Inclusion Criteria:

* Study subjects aged 22 and older.
* Subjects who sustained a Zone 2-5 flexor tendon lacerations

Exclusion Criteria:

* Subjects under the age of 22 at the time of consent
* Subjects who sustained a Zone 1 flexor tendon injury
* Subjects who have had previous surgical procedures on the injured upper extremity.
* Subjects who have metal allergies
* Ischemia, blood supply compromise, and/or inadequate wound coverage
* Prior or current infections at or near the implant site
* Conditions which tend to limit the patient's ability or willingness to restrict activities or follow directions during the healing period
* Foreign-body sensitivity
* The physical contact of the CoNextions TR Tendon Repair System with metal implants made of anything other than the implant grade of stainless steel, such as titanium, titanium alloys, cobalt chromium, or other dissimilar metals
* Surgical procedures other than for the following indication: digital flexor tendons, digital extensor tendons proximal to the metacarpophalangeal joints (Zones 6-8)
* Tendon size or surgical site access outside of specified range (Tendon Width (3.0-9.0 mm), Tendon Thickness (1.5-4.0 mm), Minimum Surgical Site Access (20 mm [10mm/side]) for the CoNextions TR Tendon Repair System

Ages: 22 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To determine the tendon failure/rupture rate of two tendon repair techniques: the CoNextions tendon repair device vs a standard of care suture repair technique. Also to determine if there are similar or different rates of complications and failures | From enrollment to end of postoperative follow up at 6-months.

SECONDARY OUTCOMES:
Time to Repair | From enrollment to end of postoperative follow up at 6-months
  The units measured will be minutes/seconds for repair
Visual Analog Pain Scale | From enrollment to end of postoperative follow up at 6-months
  Visual number scale to rate pain
Quick DASH Form | From enrollment to end of postoperative follow up at 6-months
  Assessment of symptoms and ability to perform certain activities.
Patient Satisfaction Questionnaire | From enrollment to end of postoperative follow up at 6-months
  Assessment of perceptions of technical quality, interpersonal manner, communication, financial aspects, time spent with the doctor, accessibility, and convenience, as well as overall general satisfaction.
Grip/Strength Assessment | From enrollment to end of postoperative follow up at 6-months
  Measured using a hand-held dynamometer in units of pounds/kilograms
Range of Motion Assessment | From enrollment to end of postoperative follow up at 6-months
  Measured using a goniometer and recorded in degrees.
Surgical Time | From enrollment to end of postoperative follow up at 6-months
  Total surgical time recorded in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No